CLINICAL TRIAL: NCT06915155
Title: Safety and Efficacy of the Swing-Mesh™ Implant (THT BioScience™, B. Braun™, France) in Laparoscopic-endoscopic Inguinal Hernia Repair - a Multicenter, Cohort, Prospective Observational Study.
Brief Title: Swing-Mesh™ Study (SMS).
Acronym: SMS
Status: Active, not recruiting | Type: Observational
Sponsor: Swissmed Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMS
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Inguinal Hernia
Keywords: Mesh; Groin Hernia; Hernia; TAPP; TEP; Inguinal Hernia; Minimally Invasive Surgery; Laparoscopic Hernia Repair
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Swing-Mesh™ Cohort: Patients undergoing elective laparoscopic-endoscopic inguinal hernia repair (TAPP or TEP) using the Swing-Mesh™ implant without fixation. Follow-up is conducted at 7-10 days, 30 days, 3 months, and 6 months to assess recurrence, pain, complications, and groin discomfort.
  Interventions: Device: Swing-Mesh™

INTERVENTIONS:
Device: Swing-Mesh™ — A lightweight, macroporous, three-dimensional polypropylene mesh implant developed by THT BioScience™ and distributed by B. Braun™, used in laparoscopic-endoscopic inguinal hernia repair without fixation. The mesh is designed to conform to the anatomical shape of the myopectineal orifice and is available in two sizes (15×11 cm or 16×12 cm).
  Other Names: THT BioScience mesh, 3D hernia mesh, SwingMesh, B. Braun mesh

SUMMARY:
This multicenter, prospective observational study aims to assess the safety and efficacy of the Swing-Mesh™ implant (THT BioScience™, distributed by B. Braun™, France) for laparoscopic-endoscopic inguinal hernia repair using TAPP or TEP techniques. Swing-Mesh™ is a lightweight, macroporous, three-dimensional mesh designed to conform anatomically to the myopectineal orifice without requiring fixation. Eligible adult patients undergoing elective repair will receive the implant. The primary endpoint is hernia recurrence within 6 months. Secondary endpoints include postoperative pain, groin discomfort, and early and late complications. The study will provide clinical evidence regarding the non-inferiority of this spatial, fixation-free mesh compared to standard devices in minimally invasive hernia surgery.

DETAILED DESCRIPTION:
Laparoscopic techniques such as TAPP and TEP are currently recommended as the standard approach for inguinal hernia repair due to faster recovery, reduced postoperative pain, and lower complication rates compared to open surgery.

To address the limitations of flat meshes in minimally invasive procedures, three-dimensional implants have been developed. These are better suited to the anatomical structure of the myopectineal orifice (MPO), reducing the risk of mesh migration without the need for fixation.

Swing-Mesh™ is a new lightweight, macroporous 3D implant introduced to the Polish market in 2025. Its structure is based on thermally modified polypropylene fibers, eliminating the need for rigid stabilizing rings. The implant is suitable for both right- and left-sided hernias.

The aim of this study is to assess the safety and clinical performance of Swing-Mesh™ in real-world settings. The primary endpoint is the hernia recurrence rate within 6 months. Secondary outcomes include postoperative pain, early and late complications, and patient-reported groin discomfort.

This is a prospective, multicenter, observational cohort study. Consecutive patients undergoing elective laparoscopic inguinal hernia repair will be enrolled after providing informed consent. The Swing-Mesh™ (15×11 cm or 16×12 cm) will be implanted without fixation. Selected surgical steps will be documented (photo/video), anonymized, and stored on a secure research platform.

Follow-up will be conducted at 7-10 days, 30 days, 3 months, and 6 months postoperatively. Data will be collected via structured telephone interviews or in-person visits, as needed.

ELIGIBILITY:
Inclusion Criteria:

* elective groin hernia repair
* age > 18 years
* male and female patients can participate
* eligibility for laparoendoscopic repair
* signed written informed consent

Exclusion Criteria:

* age <18 years
* emergency surgery (incarcerated hernia)
* contaminated surgical field
* recurrent hernia
* extremely large scrotal hernias with the need of other abdominal compartment syndrome (ACS) preventive procedures (botulin injection, bowel resection, preoperative progressive pneumoperitoneum - PPP)
* M3 or M3+L1-3 (EHS classification) groin hernia confirmed during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic-endoscopic inguinal hernia repair using the Swing-Mesh™ implant. The study population includes adult patients of both sexes who meet the inclusion criteria and do not have any of the specified exclusion criteria. Participants will be recruited from surgical centers in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence rate within 6 months | 6 months post-surgery
  Incidence of clinically or radiologically confirmed inguinal hernia recurrence during a 6-month follow-up period. Expected recurrence rate: 2-4%.

SECONDARY OUTCOMES:
Postoperative pain intensity (Visual Analog Scale 0-10) | 7-10 days, 30 days, 3 months, and 6 months post-surgery
  Evaluation of postoperative pain using the Visual Analog Scale (VAS) at specified time points. Chronic pain defined as pain ≥4/10 persisting beyond 3 months.
Early and late postoperative complications | Up to 6 months post-surgery
  Assessment of complications such as wound infection, hematoma, and seroma within 30 days (early) and up to 6 months (late).
Groin discomfort and foreign body sensation | 7-10 days, 30 days, 3 months, and 6 months post-surgery
  Patient-reported outcomes regarding groin discomfort and sensation of a foreign body during scheduled follow-up interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Zamkowski, MD, PhD, Study Chair — Swissmed Hospital; Maciej Śmietański, prof., Study Director — Swissmed Hospital
Locations (2):
- Poland (2):
  - Swissmed Hospital, Gdansk, Gdańsk
  - Swissmed Hospital, Gdansk

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., recurrence outcomes, VAS scores) may be shared upon reasonable request, after publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study and publication of results
Access Criteria: Requests must be made by qualified researchers with a methodologically sound proposal, subject to approval by the study investigators.

REFERENCES:
- [Result] Bittner R, Montgomery MA, Arregui E, Bansal V, Bingener J, Bisgaard T, Buhck H, Dudai M, Ferzli GS, Fitzgibbons RJ, Fortelny RH, Grimes KL, Klinge U, Kockerling F, Kumar S, Kukleta J, Lomanto D, Misra MC, Morales-Conde S, Reinpold W, Rosenberg J, Singh K, Timoney M, Weyhe D, Chowbey P; International Endohernia Society. Update of guidelines on laparoscopic (TAPP) and endoscopic (TEP) treatment of inguinal hernia (International Endohernia Society). Surg Endosc. 2015 Feb;29(2):289-321. doi: 10.1007/s00464-014-3917-8. Epub 2014 Nov 15. No abstract available. PMID 25398194
- [Result] Zamkowski M, S Mietanski M, Franczak P, Gorski D, Grabias J, Janik M, Krol A, Mitura K, Medras O, Nawacki L, Romanczuk M, Rymkiewicz P, Saluk S, Sroczynski P, Sulkowski L, Wieczorek D, Wlodarczyk M. MEsh FIxation STudy in Laparoendoscopic Repair of M3 Inguinal Hernias: Multicenter, Double-blind, Randomized Controlled Trial-MEFISTO Trial. Ann Surg. 2025 Jun 1;281(6):921-927. doi: 10.1097/SLA.0000000000006669. Epub 2025 Feb 13. PMID 39945075
- [Result] Zamkowski M, Tomaszewska A, Lubowiecka I, Karbowski K, Smietanski M. Is mesh fixation necessary in laparoendoscopic techniques for M3 inguinal defects? An experimental study. Surg Endosc. 2023 Mar;37(3):1781-1788. doi: 10.1007/s00464-022-09699-5. Epub 2022 Oct 13. PMID 36229552
- [Result] Stabilini C, van Veenendaal N, Aasvang E, Agresta F, Aufenacker T, Berrevoet F, Burgmans I, Chen D, de Beaux A, East B, Garcia-Alamino J, Henriksen N, Kockerling F, Kukleta J, Loos M, Lopez-Cano M, Lorenz R, Miserez M, Montgomery A, Morales-Conde S, Oppong C, Pawlak M, Podda M, Reinpold W, Sanders D, Sartori A, Tran HM, Verdaguer M, Wiessner R, Yeboah M, Zwaans W, Simons M. Update of the international HerniaSurge guidelines for groin hernia management. BJS Open. 2023 Sep 5;7(5):zrad080. doi: 10.1093/bjsopen/zrad080. PMID 37862616
- [Result] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835